CLINICAL TRIAL: NCT07402642
Title: Effect of Early Educational Intervention on Cardiovascular Risk Factors After Acute Coronary Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sergio Mies Padilla (Other)
Collaborators: Complejo Hospitalario Universitario Insular Materno Infantil (Other)
Responsible Party: Sponsor-Investigator, Sergio Mies Padilla, Nurse doctor in the research support unit, Servicio Canario de Salud
Organization: Servicio Canario de Salud (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2025-519-1
Record Dates: First submitted 2026-01-28; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Myocardial Infarction
Keywords: Patient Education; Secondary Prevention; Nursing Care; Self Efficacy; risk factors; Healthy Lifestyle; Cardiovascular Diseases
MeSH Terms: conditions — Myocardial Infarction; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: The study model designed for your research is defined as a quasi-experimental parallel group trial. In this design, participants are divided into two branches that progress simultaneously but independently, receiving different levels of care.
  Experimental Group (Prospective Recruitment): participants receive standard medical care plus a structured, protocol-based nursing consultation.
  Control Group (Retrospective Recruitment): participants receive standard care only, which includes the conventional cardiac rehabilitation program
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The intervention for the experimental group consists of specialized and structured nursing care provided in addition to standard medical treatment. This program is organized into four key stages: it begins with an initial contact during hospital admission to explain the objectives and assess baseline risks. Subsequently, between 7 and 10 days after discharge, a 60-minute in-person visit is conducted to perform a complete medical history and deliver adapted educational materials on heart-healthy habits. Four months after the event, a telephone reinforcement session is held to monitor treatment adherence and lifestyle changes. Finally, eight months after discharge, an in-person evaluation is carried out to measure the achievement of goals and, if necessary, refer the patient to other specialists. The entire process is supported by the use of infographics and evidence-based educational materials focused on blood pressure control, diet, exercise, and emotional health.
  Interventions: Behavioral: Motivational and Individualized Interviewing; Behavioral: Heart-Healthy Dietary Education; Behavioral: Tobacco Cessation Approach; Behavioral: Physical Activity Promotion; Behavioral: Emotional Health Management; Behavioral: Therapeutic Adherence Reinforcement; Behavioral: Self-Control Training; Behavioral: Use of Educational Resources; Other: Cardiac Rehabilitation Program
- Control Group (Active Comparator): The Control Group consists of patients who receive the standard healthcare provided by the hospital after a heart attack. These participants are recruited retrospectively using the hospital's hemodynamic service records. After discharge, they participate in the standard cardiac rehabilitation program, which typically includes 17 sessions of physical exercise and group health education. Their data is collected through a single telephone interview approximately 8 months after their heart attack to evaluate their lifestyle habits, emotional state, and clinical progress.
  Interventions: Other: Cardiac Rehabilitation Program

INTERVENTIONS:
Behavioral: Motivational and Individualized Interviewing — Used to verify the patient's understanding of their condition and to motivate behavioral changes.
  Arms: Experimental Group
Behavioral: Heart-Healthy Dietary Education — Specific counseling to improve adherence to the Mediterranean diet and address overweight or obesity
  Arms: Experimental Group
Behavioral: Tobacco Cessation Approach — Interventions aimed at increasing motivation to quit smoking and reducing nicotine dependence
  Arms: Experimental Group
Behavioral: Physical Activity Promotion — Personalized exercise recommendations tailored to the patient's clinical status
  Arms: Experimental Group
Behavioral: Emotional Health Management — Professional support to address emotional well-being, detecting potential states of anxiety or depression following the acute event.
  Arms: Experimental Group
Behavioral: Therapeutic Adherence Reinforcement — Continuous education and monitoring to ensure compliance with the prescribed pharmacological plan
  Arms: Experimental Group
Behavioral: Self-Control Training — Training the patient for autonomous monitoring of risk factors, such as blood pressure
  Arms: Experimental Group
Behavioral: Use of Educational Resources — Provision of adapted materials (infographics and written documents) to permanently reinforce healthy knowledge and behaviors
  Arms: Experimental Group
Other: Cardiac Rehabilitation Program — Upon hospital discharge, all patients are referred to a cardiac rehabilitation unit. The program consists of an average of 17 sessions focused primarily on the physical rehabilitation of the patient. Patients receive group-based health education provided by nursing professionals during these sessions.These rehabilitation sessions are typically completed within three months following the coronary event. Patients continue to receive medical and nursing attention through specialized care centers or primary care. Both groups receive optimal pharmacological treatment and general advice on cardiovascular health, including physical activity and diet.

SUMMARY:
Early Education After a Heart Attack What is the purpose of this study? The main goal is to evaluate if a special nursing education and support program helps patients who have suffered a heart attack feel more confident in managing their own health. Researchers want to see if this extra support improves how patients care for their hearts through diet, physical activity, and quitting smoking. The study compares this new nursing strategy against the standard care patients usually receive.

Who can participate? Participants must be 18 years of age or older. People who have recently had a heart attack requiring an urgent heart catheterization at the Complejo Hospitalario Universitario Insular Materno Infantil.

Exclusions: People with significant language barriers (Spanish), mental incapacity to follow recommendations, or those unable to attend in-person consultations cannot participate.

What will happen during the study? Participants will be divided into two groups: Standard Care Group (Control): These participants will receive the usual medical follow-up and standard cardiac rehabilitation sessions (an average of 17 sessions focused on exercise and group education). Special Support Group (Experimental): In addition to standard care, these participants will have a specific nursing consultation consisting of 4 scheduled visits.

These visits are a mix of in-person and telephone appointments.Nurses will provide personalized educational materials, such as infographics, and teach techniques to control blood pressure, improve diet, exercise safely, and manage emotions after a heart attack.

Duration and Follow-up Each participant will be followed for approximately 8 months. During this time, they will be asked to complete several surveys about their lifestyle.

Researchers will also review blood test results (cholesterol levels) from their medical records to track progress.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have suffered an Acute Myocardial Infarction.
* Participants must have undergone an urgent cardiac catheterization.
* Specifically, this includes patients who received coronary reperfusion strategies following the activation of the CODICAN protocol (assistance for ST-segment elevation myocardial infarction) within the study environment.

Exclusion Criteria:

* Patients with little or no knowledge of the Spanish language that prevents effective communication or reading of educational resources.
* Patients unable to understand their participation or follow health recommendations independently.
* Patients with an unfavorable clinical prognosis or those requiring hospitalization for a period exceeding established limits.
* Patients unable to attend in-person nursing consultations due to personal reasons or place of residence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2026-01-12 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Cardiac Self-Efficacy | Experimental Group: measured at two time points: baseline (during hospitalization) and 8 months (post-coronary event). Control Group: measured only at the 8-month mark post-coronary event to evaluate the level of self-efficacy after receiving standard
  His measure evaluates specific behaviors related to cardiovascular health using the Spanish-validated version of the Cardiac Self-Efficacy Scale (S-CSE). This tool consists of 12 items across three dimensions: symptom control, disease control, and activity maintenance. Each item is rated on a 7-point Likert scale (1 = not at all confident, 7 = completely confident). Total scores range from 12 to 84, where higher scores indicate better self-efficacy

SECONDARY OUTCOMES:
Adherence to the Mediterranean Diet | Experimental Group: baseline and 8 months Control Group: 8 months only
  Measured using the MEDAS questionnaire (14 items). Higher scores indicate greater adherence to a heart-healthy diet
Nicotine Dependence | Experimental Group: baseline and 8 months Control Group: 8 months only
  Assessed using the Fagerström Test (6 items). Scores range from 0 to 10, where greater than or equal to 7 indicates high dependence
Motivation to Quit Smoking | Experimental Group: Baseline and 8 months . Control Group: 8 months only.
  Evaluated through the Richmond Test (4 items). Scores range from 0 to 10; scores between 8-10 indicate high motivation.
Physical Activity Level | Experimental Group: Baseline and 8 months Control Group: 8 months only.
  Measured using the International Physical Activity Questionnaire (IPAQ). It categorizes patients into high, moderate, or low activity levels based on METs.
Affective State (Anxiety and Depression) | Experimental Group: Baseline and 8 months Control Group: 8 months only
  Determined using the Goldberg Scale. It consists of two subscales (anxiety mayor o igual a 4 and depression greater than or equal to 2) to detect psychological distress
Lipid Profile | Experimental Group: Baseline and 8 months Control Group: 8 months only
  Clinical data collection of total cholesterol, LDL, HDL, and triglycerides from medical records
Cardiac Rehabilitation Adherence | 8 months (for both groups)
  Exploration of patient inclusion, adherence (number of sessions attended), and group education received

CONTACTS AND LOCATIONS:
Locations (1):
- Complejo Hospitalario Universitario Insular Materno Infantil de Gran Canaria, Las Palmas de Gran Canaria, Las Palmas, Spain

IPD SHARING:
Plan to Share IPD: No
Currently, there is no plan to share individual participant data (IPD) with external researchers or public platforms. According to the protocol, the collected data will be used exclusively for the research purposes of this specific study, and only the research team will have access to the anonymized database. Patient privacy is protected by current regulations (Spanish Organic Law 3/2018), ensuring that information is treated confidentially and securely within the hospital environment.